CLINICAL TRIAL: NCT06013098
Title: Effects of Different Oxygen Concentrations on Pulmonary Complications in Patients Undergoing Radical Resection of Esophageal Cancer
Acronym: DOICA-E
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Wenfei Tan, Professor, China Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20230724-2
Record Dates: First submitted 2023-08-22; First posted 2023-08-28 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Atelectasis, Postoperative
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: 30% Oxygen (Experimental): Before anesthesia induction, the participants inhaled pure oxygen through the mask for 5 minuets. After successful anesthesia induction, FiO2 will be adjusted to 60% in one lung ventilation and 30% FIO2 in both lungs ventilation, and the total gas flow rate will be set at 2L/min. All patients will be performed via the lung protective ventilation strategy. The respiratory parameters are VT: 6-8ml/kg, PEEP: 6-8 cm H2O, RR: 1:2. Manual lung recruitment maneuvers will be performed after tracheal intubation and before tracheal extubation, however when intraoperative oxygen saturation is less than 92% the manual lung recruitment maneuver will be done too. Arterial blood will be collected for blood gas analysis. Patients in both groups will be extubation the operating room and then sent to the PACU. patients should transfer to 60% Oxygen group if intraoperative oxygen saturation less than 85%.
  Interventions: Drug: 30%Oxygen
- Experimental: 60% Oxygen (Placebo Comparator): Before anesthesia induction, the participants inhaled pure oxygen through the mask for 5 minutes. After successful anesthesia induction, FiO2 will be adjusted to 100% in one lung ventilation and 60% FIO2 in both lungs ventilation, and the total gas flow rate will be set at 2L/min. All patients will be performed via the lung protective ventilation strategy. The respiratory parameters are VT: 6-8ml/kg, PEEP: 6-8 cm H2O, RR: 1:2. Manual lung recruitment maneuvers will be performed after tracheal intubation and before tracheal extubation, however when intraoperative oxygen saturation is less than 92% the manual lung recruitment maneuver will be done too. Arterial blood will be collected for blood gas analysis. Patients in both groups will be extubation the operating room and then sent to the PACU.
  Interventions: Drug: 60%Oxygen

INTERVENTIONS:
Drug: 30%Oxygen — 60%FiO2 in one lung ventilation and 30% FIO2 in both lungs ventilation
  Arms: Experimental: 30% Oxygen
Drug: 60%Oxygen — 100%FiO2 in one lung ventilation and 60% FIO2 in both lungs ventilation
  Arms: Experimental: 60% Oxygen

SUMMARY:
Radical operation of esophageal cancer is complicated and traumatic, and ventilation with one lung in lateral position and ventilation with both lungs after supine position requires long-term tracheal intubation and ventilator-assisted ventilation, and the incidence of postoperative pulmonary complications is high.

DETAILED DESCRIPTION:
Therefore, we should explore the most appropriate lung protection ventilation strategy to reduce the occurrence of pulmonary complications. The recommended standard of international expert group on lung protective ventilation strategy points out that the lowest concentration of oxygen (≤40%) should be inhaled as much as possible during mechanical ventilation to maintain normal blood oxygen level (SpO2≥94%). If the mixed gas with low inhaled oxygen concentration can achieve ideal oxygen saturation and arterial oxygen partial pressure, it may reduce the postoperative pulmonary complications of the subjects. However, there are few reports on the influence of different oxygen concentrations on pulmonary complications in patients undergoing radical resection of esophageal cancer. This study intends to explore the influence of different oxygen concentrations on pulmonary complications in patients undergoing radical resection of esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* American Association of Anesthesiologists (ASA) patients with I-II physical condition;
* Patients with preoperative partial pressure of blood gas and oxygen greater than 80mmHg who were scheduled for elective esophageal cancer surgery were operated in the right lateral position first and then in the supine position.

Exclusion Criteria:

* there is a history of acute lung injury with acute respiratory distress syndrome within three months;
* Heart failure (classified by new york Heart Association) is greater than grade IV,
* there is a serious liver and kidney dysfunction (children with grade B or C liver failure, glomerular filtration rate < 30 ml/min);
* Body mass index > 30kg/m2；
* coagulation dysfunction;
* Operation time exceeds 10h
* The amount of bleeding is more than 800ml, and the total fluid volume is more than 3000ml.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-06 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
the occurrence of atelectasis | On the operating room within 40 minutes after awakening
  The primary outcome is the occurrence of atelectasis scanned by computerized tomography in the operating room within 40 minutes after awakening

SECONDARY OUTCOMES:
oxygenation index | On the operating room within 40 minutes after awakening
  The secondary outcome is the comparison of the oxygenation index between the two groups, which is calculated and compared from the results of intraoperative blood gas analysis

CONTACTS AND LOCATIONS:
Locations (1):
- the First Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided